CLINICAL TRIAL: NCT02515227
Title: A Trial to Evaluate the Safety, Immunogenicity, and Clinical Activity of a Helper Peptide Vaccine Plus PD-1 Blockade
Brief Title: Safety Study of a Helper Peptide Vaccine Plus Pembrolizumab
Acronym: Mel64
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Craig L Slingluff, Jr (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Craig L Slingluff, Jr, Director, Human Immune Therapy Center, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18174; R01CA178846 (NIH)
Record Dates: First submitted 2015-07-30; First posted 2015-08-04 (Estimated); Results first posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Melanoma
Keywords: peptide; vaccine; Montanide ISA-51; pembrolizumab; PD-1; KEYTRUDA
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 6MHP (6 Melanoma helper peptide) vaccine + Pembrolizumab (Experimental): 6MHP (200 mcg each peptide) will be administered intradermally and subcutaneously on days 1, 8, 15, 43, 64, and 85. Pembrolizumab (200 mg) will be administered intravenously every 3 weeks for up to 2 years, beginning on day 1.
  Interventions: Biological: 6MHP; Drug: Pembrolizumab

INTERVENTIONS:
Biological: 6MHP — 6 melanoma helper vaccine comprised of 6 class II MHC-restricted helper peptides
  Other Names: 6 melanoma helper peptide vaccine
Drug: Pembrolizumab — Humanized monoclonal antibody (mAb) specific for PD-1.
  Other Names: KEYTRUDA; MK-3475

SUMMARY:
This study evaluates whether it is safe to administer a peptide vaccine in combination with pembrolizumab. This study will also evaluate the effects of the combination of the peptide vaccine and pembrolizumab on the immune system. The investigators will monitor these effects by performing tests in the laboratory on participants' blood, a lymph node, and tumor samples.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with unresectable American Joint Committee on Cancer (AJCC) stage IIIB or stage IIIC melanoma, or stage IV metastatic melanoma that have clinical or radiological evidence of disease. Subjects may have had cutaneous, uveal, mucosal primary melanoma, or an unknown primary melanoma. Staging must be confirmed by cytological or histological examination. Staging of cutaneous melanoma will be based on the revised AJCC staging system
2. Ability to provide written informed consent/assent for the trial.
3. ≥18 years of age
4. A subject may be naïve for immunotherapy agents or have received interferon-alpha, ipilimumab or other cytotoxic T lymphocyte antigen (CTLA)-4 antibody, Programmed death-1 (PD-1) antibody (or anti-PD-L1 antibody), interleukin-2, or prior cancer vaccines other than the 6MHP vaccine. Patients who have received a PD-1/PD-L1 antibody may be enrolled in either of the following settings:

   1. A patient who has experienced progression of melanoma during that therapy or after having completed that therapy,
   2. A patient who fails to experience an objective clinical response (partial response or complete response by RECIST 1.1 criteria) after either 12 weeks of continuous anti-PD1 antibody or anti-CTLA4/anti-PD1 combination therapy, and is a candidate to receive pembrolizumab therapy
5. Measurable disease based on RECIST 1.1.

   Subjects will be required to have radiological studies to define radiologically evident disease. Required studies include:
   * Chest CT scan,
   * Abdominal and pelvic CT scan, and
   * Head CT scan or MRI Positron emission tomography (PET)/CT fusion scan may replace scans of the chest, abdomen, and pelvis.
6. Subjects who have metastatic melanoma available for biopsy pretreatment and on day 22 must consent to having those biopsies. These metastases may be in nodes, skin, soft tissue, liver, or other sites that can be accessed safely by needle biopsy, incisional or excisional biopsy, with or without image guidance. The lesions to be biopsied must be specified at study enrollment and not included as target lesions for RECIST calculations. In instances where disease that is accessible to biopsy is limited, archival tissue specimens collected after a subject's last systemic therapy may be used for baseline measures.

   Subjects must have measurable disease in addition to the lesion(s) to be biopsied.
7. Subjects who have had brain metastases will be eligible if all of the following are true:

   * Each brain metastasis must have been completely removed by surgery or each unresected brain metastasis must have been treated with stereotactic radiosurgery.
   * There has been no evident growth of any brain metastasis since the most recent treatment
   * No brain metastasis is > 2 cm in diameter at the time of registration.
   * Neurologic symptoms have returned to baseline,
   * There is no evidence of new or enlarging brain metastases,
   * Subjects are not using steroids for at least 7 days prior to registration.
8. The most recent surgical resections or gamma-knife therapy for malignant melanoma must have been completed ≥ 1 week prior to registration.
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
10. Adequate organ function.
11. Two intact (undissected) axillary and/or inguinal lymph node basins.

Exclusion Criteria

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
2. Is currently receiving Interferon (e.g. Intron-A®), growth factors (e.g. Procrit®, Aranesp®, Neulasta®), or interleukins (e.g. Proleukin®), or has received these agents within 4 weeks of the first dose of treatment.
3. Is currently receiving nitrosureas or has received this therapy within the preceding 6 weeks of first dose of treatment.
4. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment with the following exceptions (which are permitted):

   * replacement steroid doses in patients with adrenal or pituitary insufficiency
   * Intra-articular steroid injections
   * Inhaled steroids (e.g.: Advair®, Flovent®, Azmacort®) at low doses (less than 500 mcg fluticasone per day, or equivalent)
   * Topical and nasal corticosteroids
   * Non-steroidal anti-inflammatory drugs
5. Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e. ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or external beam radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include carcinoma in situ of the breast (DCIS or LCIS), basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
9. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Exceptions to this criterion include:

   * Subjects with vitiligo or other depigmenting illness.
   * Resolved childhood asthma/atopy
   * Intermittent use of bronchodilators or local steroid injections
   * Hypothyroidism stable on hormone replacement or Sjogren's syndrome
   * The presence of laboratory evidence of autoimmune disease (e.g. positive ANA titer) without symptoms
   * Mild arthritis requiring NSAID medications
10. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
15. Is HIV positive or has evidence of active Hepatitis C virus (testing to be done within 6 months of study entry) or active Hepatitis B virus.
16. Has received a live vaccine or allergy desensitization injections within 30 days prior to the first dose of trial treatment.
17. Has known or suspected allergies to any component of the vaccine.
18. Has been vaccinated previously with any of the synthetic peptides included in this protocol.
19. Is classified according to the New York Heart Association classification as having Class III or IV heart disease (Appendix 12.5).
20. Has uncontrolled diabetes, defined as having a HGBA1C > 7.5%.
21. Has a body weight < 110 pounds (without clothes) at enrollment, due to the amount and frequency with which blood will be drawn.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig L. Slingluff, Jr., MD, Study Director — University of Virginia
Locations (1):
- University of Virginia Cancer Center, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were all enrolled at the University of Virginia Cancer Center and were treated as outpatients.
  The study opened to enrollment 11/19/2015. The first participant was enrolled 10/6/2016. The first participant's first treatment was 10/10/2016. The last participant was enrolled 6/26/2019.
Groups:
- 6MHP + Pembrolizumab (PD-1 Antibody-naive Cohort): Participants who had not previously received a PD-1 or PD-L1 antibody were eligible for this cohort.
  They received 6MHP vaccine (200 mcg each peptide) emulsified in Montanide ISA-51 adjuvant and administered intradermally and subcutaneously on days 1, 8, 15, 43, 64, and 85. Pembrolizumab (200 mg) was administered intravenously every 3 weeks for up to 2 years, beginning on day 1.
  6MHP: 6 melanoma helper vaccine comprised of 6 class II MHC-restricted helper peptides
  Pembrolizumab: Humanized monoclonal antibody (mAb) specific for PD-1.
- 6MHP + Pembrolizumab (PD-1 Antibody-experienced Cohort): Participants who had previously received a PD-1 or PD-L1 antibody were eligible for this cohort.
  They received 6MHP vaccine (200 mcg each peptide) emulsified in Montanide ISA-51 adjuvant and administered intradermally and subcutaneously on days 1, 8, 15, 43, 64, and 85. Pembrolizumab (200 mg) was administered intravenously every 3 weeks for up to 2 years, beginning on day 1.
  6MHP: 6 melanoma helper vaccine comprised of 6 class II MHC-restricted helper peptides
  Pembrolizumab: Humanized monoclonal antibody (mAb) specific for PD-1.
Period: Overall Study
Arm/Group | 6MHP + Pembrolizumab (PD-1 Antibody-naive Cohort) | 6MHP + Pembrolizumab (PD-1 Antibody-experienced Cohort)
Started | 6 | 16
Received at Least 1 Vaccine | 6 | 16
Completed (This milestone reflects receipt of all 6 vaccines and remaining on study to week 13 at least.) | 4 | 5
Not Completed | 2 | 11
Not completed — Adverse Event | 0 | 2
Not completed — Progressive disease | 2 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 6MHP + Pembrolizumab (PD-1 Antibody-naive Cohort) | 6MHP + Pembrolizumab (PD-1 Antibody-experienced Cohort) | Total
Number analyzed (Participants) | 6 | 16 | 22
Age, Customized [Median (Full Range); unit: years]
  Age at enrollment | 71.5 [44 to 81] | 62.5 [36 to 75] | 63 [36 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 8 | 9
  Male | 5 | 8 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race at Enrollment: Caucasian/White: non-Hispanic | 6 | 15 | 21
  Race at Enrollment: African-American/Black: non-Hispanic | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 16 | 22
ECOG Performance Status [Count of Participants; unit: Participants] — This measure of performance status refers to a scale from 0 to 5. Grade 0 refers to normal health with full activity and normal activity performance. Grade 1 refers to the status where individuals are restricted in strenuous activity but they are ambulatory and able to perform light or sedentary work. Eligibility for this trial required ECOG performance status of 0 to 1.
  Participants
    0 | 4 | 9 | 13
    1 | 2 | 7 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities.
Description: Number of participants with dose-limiting toxicities on treatment with combination of pembrolizumab and 6MHP.
Time Frame: 30 days after the last administration of study drug.
Population: DLT was defined as unexpected adverse event (AE) at least possibly related to treatment, and, for 6MHP, grade ≥3 hematological or non-hematological toxicity, except that vaccine site ulcers were considered DLTs if ulcer >2cm, required antibiotics or debridement; and for pembrolizumab, required permanent discontinuation per specified guidelines. Also considered DLTs were selected grade ≥2 ocular AEs, and AEs that led to stopping treatment even if they did not meet prespecified DLT criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | 6MHP + Pembrolizumab (PD-1 Antibody-naive Cohort) | 6MHP + Pembrolizumab (PD-1 Antibody-experienced Cohort)
Number analyzed (Participants) | 6 | 16
Participants | 0 | 3

2. Primary Outcome: CD4+ T Cell Responses Detected in the Peripheral Blood or Vaccine-draining Lymph Node (Sentinel Immunized Node).
Description: Circulating CD4+ T cell responses to 6MHP peptides were assessed using IFN-γ ELISpot assays directly ex vivo for peripheral blood mononuclear cells (PBMC) and sentinel immunized node (SIN) lymphocytes. For each sample, the following definitions applied: Nvax=number of T cells responding to vaccine peptide; Nneg=number of T cells responding to maximum negative control; Rvax=Nvax/Nneg. For PBMC, a participant was considered to have a T-cell response (Rsp) if all the following were true: (1) Nvax exceeded Nneg by ≥ 20/100,000 CD4+ cells (0.02%), (2) (Nvax-1 SD)≥(Nneg+1 SD), (3) Rvax ≥2×, and (4) Rvax postvaccine ≥2x Rvax prevaccine. Criteria for CD4+ Rsp in a SIN included criterion (1-3). A high durable T cell response (hdRsp) required a 5× increase above baseline in any two or more time points (through day 85), and a durable immune response (dRsp) required only a 2× increase over background. A response in either PBMC or in SIN is considered a response for this endpoint.
Time Frame: through week 104
Measure: Count of Participants; unit: Participants
Arm/Group | 6MHP + Pembrolizumab (PD-1 Antibody-naive Cohort) | 6MHP + Pembrolizumab (PD-1 Antibody-experienced Cohort)
Number analyzed (Participants) | 6 | 16
Participants
  CD4 T cell response (Rsp): T cell response | 4 | 2
  CD4 T cell response (Rsp): No T cell response | 2 | 14
  CD4 high durable T cell response (hdRsp): T cell response | 1 | 0
  CD4 high durable T cell response (hdRsp): No T cell response | 5 | 16
  CD4 durable T cell response (dRsp): T cell response | 1 | 1
  CD4 durable T cell response (dRsp): No T cell response | 5 | 15

3. Secondary Outcome: Number of T Cells in the Tumor Microenvironment
Description: Evaluation of tumor infiltration by T cells.Tumor biopsies were obtained pretreatment and day 22 for 12 participants and were evaluated with multiplex immunofluorescence histology (mIFH). CD8+ T cell data were evaluated. CD4+ T cells were not reported because of technical challenges with that antibody. These 12 participants with evaluable tumor samples included 3 on the PD-1 antibody-naive cohort, and 9 on the antibody-experienced cohort.
Time Frame: up to day 22
Measure: Median (Inter-Quartile Range); unit: cells per mm^2 tumor
Groups:
- 6MHP + Pembrolizumab (PD-1 Antibody-naive Cohort): Participants received 6MHP vaccine (200 mcg each peptide) emulsified in Montanide ISA-51 adjuvant and administered intradermally and subcutaneously on days 1, 8, 15, 43, 64, and 85. Pembrolizumab (200 mg) was administered intravenously every 3 weeks for up to 2 years, beginning on day 1.
  6MHP: 6 melanoma helper vaccine comprised of 6 class II MHC-restricted helper peptides
  Pembrolizumab: Humanized monoclonal antibody (mAb) specific for PD-1.
- 6MHP + Pembrolizumab (PD-1-experienced Cohort): Participants who had previously received a PD-1 or PD-L1 antibody were eligible for this cohort.
  They received 6MHP vaccine (200 mcg each peptide) emulsified in Montanide ISA-51 adjuvant and administered intradermally and subcutaneously on days 1, 8, 15, 43, 64, and 85. Pembrolizumab (200 mg) was administered intravenously every 3 weeks for up to 2 years, beginning on day 1.
  6MHP: 6 melanoma helper vaccine comprised of 6 class II MHC-restricted helper peptides
  Pembrolizumab: Humanized monoclonal antibody (mAb) specific for PD-1.
Arm/Group | 6MHP + Pembrolizumab (PD-1 Antibody-naive Cohort) | 6MHP + Pembrolizumab (PD-1-experienced Cohort)
Number analyzed (Participants) | 3 | 9
cells per mm^2 tumor
  CD8 T cells per mm^2 in day 0 tumor | 28.7 [16.7 to 324.9] | 125.5 [18.9 to 267.1]
  CD8+ T cells per mm^2 in day 22 tumor | 259.1 [179.6 to 396.33] | 164.7 [63.1 to 585.4]

4. Secondary Outcome: Level of Th1-dominant Immune Signatures in the Tumor Microenvironment
Description: Evaluation of cytokine profile for CD4+ T cells in tumor microenvironment. Data for this outcome have not been collected due to completion of funding for this study.
Time Frame: up to day 22
Population: Immune signature data have not been collected from the tumor microenvironment.
Arm/Group | 6MHP + Pembrolizumab (PD-1 Antibody-naive Cohort) | 6MHP + Pembrolizumab (PD-1 Antibody-experienced Cohort)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of CD8+ T Cell Responses to Defined Melanoma Antigens
Description: Evaluation of epitope-spreading through the measurement of the induction of CD8+ T cell responses to defined melanoma antigens.
Time Frame: up to week 104
Population: Due to completion of funding for this study, data have not been collected to assess epitope-spreading through the measurement of the induction of CD8+ T cell responses to defined melanoma antigens.
Arm/Group | 6MHP + Pembrolizumab (PD-1 Antibody-naive Cohort) | 6MHP + Pembrolizumab (PD-1 Antibody-experienced Cohort)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Amount of IgG Antibody Specific for 6MHP as Measured in the Blood and the Sentinel Immunized Node
Description: Evaluation of antibody responses to 6MHP
Time Frame: up to week 104
Population: Antibody responses to 6MHP have not been measured, due to completion of funding for this trial.
Arm/Group | 6MHP + Pembrolizumab (PD-1 Antibody-naive Cohort) | 6MHP + Pembrolizumab (PD-1 Antibody-experienced Cohort)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events and dose-limiting toxicities (DLTs) were monitored up to 30 days after the last study treatment.
Arm/Group | 6MHP + Pembrolizumab (PD-1 Antibody-naive Cohort) | 6MHP + Pembrolizumab (PD-1 Antibody-experienced Cohort)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/16
Other Adverse Events (participants affected / at risk) | 6/6 | 16/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 6MHP + Pembrolizumab (PD-1 Antibody-naive Cohort) (N=6) | 6MHP + Pembrolizumab (PD-1 Antibody-experienced Cohort) (N=16)
Anemia (Blood and lymphatic system disorders) | 1 | 8
Adrenal Insufficiency (Endocrine disorders) | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 5
Chills (General disorders) | 1 | 2
Fatigue (General disorders) | 4 | 14
Fever (General disorders) | 3 | 3
Flu-like symptoms (General disorders) | 1 | 1
Injection site reaction (General disorders) | 6 | 14
Pain (General disorders) | 0 | 2
Bruising (Injury, poisoning and procedural complications) | 2 | 3
Alanine Aminotransferase increased (Investigations) | 0 | 2
Alkaline phosphatase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 5
Creatinine increased (Investigations) | 0 | 2
Lymphocyte count decreased (Investigations) | 2 | 4
Anorexia (Metabolism and nutrition disorders) | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Myalgia (Metabolism and nutrition disorders) | 2 | 2
Headache (Nervous system disorders) | 1 | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 4
Pruritis (Skin and subcutaneous tissue disorders) | 3 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 3
Skin induration (Skin and subcutaneous tissue disorders) | 5 | 11
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/27/NCT02515227/Prot_SAP_ICF_000.pdf